CLINICAL TRIAL: NCT00461747
Title: A National, Open-Label, Multicenter, Randomized, Comparative Phase III Study of Induction Treatment With VBMCP-VBAD/Velcade Versus Thalidomide / Dexamethasone Versus Velcade / Thalidomide / Dexamethasone Followed by High Dose Intensive Therapy With Autologous Hemopoietic Stem Cell Support and Maintenance Treatment With Interferon-a Versus Thalidomide Versus Thalidomide / Velcade in Untreated Patients With Multiple Myeloma Less Than 65 Yrs Old
Brief Title: GEM05 for Patients With Multiple Myeloma Under 65 Years
Acronym: GEM05MENOS65
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: pethema, pethema
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-001110-41
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Multiple Myeloma
Keywords: Untreated; Transplant; Younger
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Dexamethasone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Four alternating cycles of VBMCP/VBAD + Velcade VBMCP: Vincristine, 0,03 mg/Kg (iv) day 1, BCNU, 0,5 mg/Kg iv day 1, Cyclophosphamide, 10 mg/Kg iv day 1, Melfalán, 0,25 mg/Kg oral days 1 to 4 Prednisone, 1 mg/Kg oral days 1 to 4; 0,5 mg/Kg oral days 5 to 8 and 0,25 mg/Kg oral days 9 to 12.
  VBAD : Vincristine, 1mg via iv day 1, BCNU, 30 mg/m2 iv day 1, Adriamycine, 40mg/m2 iv day 1 Dexamethasone, 40 mg oral days 1 to 4, 9 to 12 and 17 to 20. The interval between VBMCP and VBAD is 5 weeks and between VBAD and VBMCP is 4 weeks. The patients will received two cycles of VBMCP and two cycles of VBAD. After 4 weeks of last cycle of VBAD, patients will received two cycles of Velcade, 1,3 mg/ m2 iv twice a week (days 1, 4, 8 and 11), followed by 10 days without treatment
  Interventions: Drug: VBMCP/VBAD/Velcade
- B (Experimental): Six cycles of 4 weeks of Thalidomide/Dexamethasone. Thalidomide day 1, cycle 1 (50 mg/day v.o). If toxicity < grade 2, dose will be 100 mg/day on day 15, cycle 1 and 200 mg/day on day 1, cycle 2.
  Dexamethasone:40 mg/day v.o.days 1 to 4 and 9 to 12, with a period without treatment of 16 days
  Interventions: Drug: Thalidomide/Dexamethasone
- C (Experimental): Thalidomide: day 1 cycle 1 (50 mg/day).If toxicity is < grade 2, the dose will be increased (100 mg/day) at day 15 cycle 1 and (200 mg de Thalidomide) at day 1 cycle 2.
  Dexamethasone: 40 mg/day v.o days 1 to 4 and 8 to 11, with a period without treatment of 17 days.
  Velcade: 1,3 mg/m2 iv twice a week (days 1, 4, 8 and 11) with a period without treatment of 17 days.
  Interventions: Drug: Velcade/Thalidomide/Dexamethasone

INTERVENTIONS:
Drug: VBMCP/VBAD/Velcade — VBMCP: Vincristine, 0,03 mg/Kg (iv) day 1, BCNU, 0,5 mg/Kg iv day 1, Cyclophosphamide, 10 mg/Kg iv day 1, Melfalan, 0,25 mg/Kg oral days 1 to 4 Prednisone, 1 mg/Kg oral days 1 to 4; 0,5 mg/Kg oral days 5 to 8 and 0,25 mg/Kg oral days 9 to 12.
  VBAD : Vincristine, 1mg via iv day 1, BCNU, 30 mg/m2 iv day 1, Adriamycine, 40mg/m2 iv day 1 Dexamethasone, 40 mg oral days 1 to 4, 9 to 12 and 17 to 20.
  Arms: A
Drug: Thalidomide/Dexamethasone — Thalidomide day 1, cycle 1 (50 mg/day v.o). If toxicity < grade 2, dose will be 100 mg/day on day 15, cycle 1 and 200 mg/day on day 1, cycle 2.
  Dexamethasone:40 mg/day v.o.days 1 to 4 and 9 to 12, with a period without treatment of 16 days
  Arms: B
Drug: Velcade/Thalidomide/Dexamethasone — Thalidomide: day 1 cycle 1 (50 mg/day).If toxicity is < grade 2, the dose increased (100 mg/day) at day 15 cycle 1 and (200 mg de Thalidomide) at day 1 cycle 2.
  Dexamethasone: 40 mg/day v.o days 1 to 4 and 8 to 11, with a period without treatment of 17 days.
  Velcade: 1,3 mg/m2 iv twice a week (days 1, 4, 8 and 11) with a period without treatment of 17 days
  Arms: C

SUMMARY:
The primary objective is to compare safety and efficacy of three induction treatments: VBMCP-VBAD / Velcade versus Thalidomide / Dexamethasone versus Velcade / Thalidomide / Dexamethasone. The second one is to evaluate the ability of stem cell mobilization after the treatments in order to do an autologous transplant. Otherwise this study wants to compare the safety and efficacy of the maintenance treatments: Interferón a-2b versus Thalidomide versus Thalidomide/Velcade.

DETAILED DESCRIPTION:
A total of up to 390 patients ≤ 65 years old diagnosed of Multiple Myeloma with symptomatic disease and that have not received previous chemotherapy for MM will be included.

Patients will be evaluated at scheduled visits in up to three study periods: Pre-treatment, Treatment and Follow up.

The Pre-treatment includes Screening and baseline visits. After providing informed consent, patients will be evaluated for study eligibility and then Patients will be randomized (1:1:1) to receive VBMCP-VBAD+Velcade (Group A) or Thalidomide+Dexamethasone (Group B) or Thalidomide+Dexamethasone+Velcade (Group C). All of them will received the induction treatment up to 24 weeks.

After 4 weeks, without progression or unacceptable toxicity, There will be stem cell mobilization to do an autologous transplant. Three months after transplant, patients will be again randomized (1:1:1) to receive maintenance treatment: Interferon-a (Group M1) or Thalidomide (Group M2) or Thalidomide+Velcade (Group M3) during three years.

Once the treatment period has finished a follow up will be carry out. During this period we will evaluated response, progression-free survival and global survival every three months.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to comply with the protocol requirements
2. Must voluntary sign the informed consent before performance of any study-related procedure not part of normal medical care,
3. Age <65 years and possibly to do an autologous transplant.
4. Patient recently diagnosed with symptomatic Multiple Myeloma who has not received any previous chemotherapy treatment for Multiple Myeloma.
5. Patient has a measurable disease defined as quantifiable serum monoclonal protein value and, where applicable, urine Light-chain excretion of ≥ 200 mg/24 hours.
6. ECOG < 2.
7. El patient has a life-expectancy > 3 months.
8. Patient has the following laboratory values before beginning induction treatment:

   1. Platelet count ≥ 50000/mm3, hemoglobin ≥ 8 g/dl and absolute neutrophil count ≥ 1000/mm3. Lower values are allowed if they are due to marrow infiltration.
   2. Corrected serum calcium <14mg/dl.
   3. Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal.
   4. Alanine transaminase (ALT): ): ≤ 2.5 x the upper limit of normal.
   5. Total bilirubin: ≤1.5 x the upper limit of normal.
   6. Serum creatinine ≤ 2 mg/dl.
9. For Patients included in Thalidomide branches: women of childbearing age must not have sex unless they use two anticonceptive methods beginning 4 weeks before the first dose, during all the study until 4 weeks after the last one.

Exclusion Criteria:

1. Non-secretor Myeloma.
2. Patients previously received treatment to Multiple Myeloma, except steroids doses for urgency or bisphosphonates or radiotherapy before beginning treatment.
3. Patients with < Grade 2 peripheral neuropathy within 14 days before enrolment.
4. Patient had major surgery within 4 weeks before enrolment.
5. Patient has hypersensitivity to bortezomib, boron or mannitol or Thalidomide.
6. Patient has received other investigational drugs within 30 days before enrolment.
7. Patient is known to be seropositive for the human immunodeficiency virus (HIV), Hepatitis B surface antigen-positive or active hepatitis C infection.
8. Patient had a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
9. Patient is enrolled in another clinical research study and/or is receiving an investigational agent for any reason.
10. Pregnancy or breast-feed women.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is to compare safety and efficacy of three induction treatments: VBMCP-VBAD / Velcade versus Thalidomide / Dexamethasone versus Velcade / Thalidomide / Dexamethasone. | 2 years

SECONDARY OUTCOMES:
Evaluate the ability of stem cell mobilization after the treatments in order to do an autologous transplant. Otherwise this study wants to compare the safety and efficacy of the maintenance treatments: Interferón a-2b versus Thalidomide | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bladé Joan, Dr, Principal Investigator — Hospital Clinic of Barcelona
Locations (79):
- Spain (79):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital Royo Villanova, Zaragoza, Aragon
  - Hospital Ntra. Sra. Sonsoles, Ávila, Avila
  - Xarxa assistencial de Manresa, Manresa, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital general de Castellón, Castelló, Castellón
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Oviedo
  - Hospital del Río Carrión, Palencia, Palencia
  - Hospital Joan XXIII, Tarragona, Tarragona
  - Hospital Clínic, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Fundación Hospital Alcorcón, Alcorcón
  - Hospital Regional Universitario Infanta Cristina, Badajoz
  - Hospital de Badalona Germans Trias i Pujol, Badalona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Basurtuko Ospitalea, Bilbao
  - Hospital de Cruces, Bilbao
  - Hospital Virgen del Puerto, Cáceres
  - Hospital Nuestra Señora de Alarcos, Ciudad Real
  - Hospital Virgen de la Luz, Cuenca
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital General de Elda, Elda
  - Hospital Universitario de Getafe, Getafe
  - Hospital General de Guadalajara, Guadalajara
  - Hospital de San Jorge, Huesca
  - Hospital General de Lanzarote, Lanzarote
  - Complejo Hospitalario León, León
  - Complexo Hospitalario Xeral-Calde, Lugo
  - Clínica Moncloa, Madrid
  - Clínica Puerta de Hierro, Madrid
  - Clínica Rúber, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Central de la Defensa, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Fundación Hospital Sant Joan de Déu de Martorell, Martorell
  - Hospital de Mérida, Mérida
  - Hospital General Morales Meseguer, Murcia
  - Hospital Santa María del Rosell, Murcia
  - Hospital Virgen del Castillo de Yecla, Murcia
  - Hospital de Gran Canaria Doctor Negrín, Palma de Gran Canaria
  - Complejo Asistencial Son Dureta, Palma de Mallorca
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Verge del Toro, Palma de Mallorca
  - Hospital de Navarra, Pamplona
  - Hospital Virgen del Camino, Pamplona
  - Complejo Hospitalario de Pontevedra_Hospital Montecelo, Pontevedra
  - Complejo Hospitalario de Pontevedra_Hospital Provincial, Pontevedra
  - Hospital de Sagunto, Sagunto
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital San Pedro de Alcántara, San Pedro
  - Clínica Sant Camil, Sant Pere de Ribes
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Hospital Nuestra Señora del Prado, Toledo
  - Hospital Virgen de la Salud, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Dr. Peset, Valencia
  - Hospital Francesc de Borja, Valencia
  - Hospital General Básico de la Defensa, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Comarcal de Vinaros, Vinaròs
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital de Galdakao, Vizcaya
  - Hospital Virgen de la Concha, Zamora
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Background] Greenlee RT, Murray T, Bolden S, Wingo PA. Cancer statistics, 2000. CA Cancer J Clin. 2000 Jan-Feb;50(1):7-33. doi: 10.3322/canjclin.50.1.7. PMID 10735013
- [Background] 2. Longo D. Plasma cell disorders. In : Fauce A, et al. Ed. Harrison's Principles of Internal Medicine. 14th Ed. New York, New York: Mc Graw-Hill; 1998: 712-718
- [Background] Raje N, Anderson K. Thalidomide--a revival story. N Engl J Med. 1999 Nov 18;341(21):1606-9. doi: 10.1056/NEJM199911183412110. No abstract available. PMID 10564693
- [Background] Oken MM. Management of Myeloma: Current and Future Approaches. Cancer Control. 1998 May;5(3):218-225. doi: 10.1177/107327489800500302. PMID 10761055
- [Background] Holland JR, Hosley H, Scharlau C, Carbone PP, Frei E 3rd, Brindley CO, Hall TC, Shnider BI, Gold GL, Lasagna L, Owens AH Jr, Miller SP. A controlled trial of urethane treatment in multiple myeloma. Blood. 1966 Mar;27(3):328-42. No abstract available. PMID 5933438
- [Background] Alexanian R, Haut A, Khan AU, Lane M, McKelvey EM, Migliore PJ, Stuckey WJ Jr, Wilson HE. Treatment for multiple myeloma. Combination chemotherapy with different melphalan dose regimens. JAMA. 1969 Jun 2;208(9):1680-5. doi: 10.1001/jama.208.9.1680. No abstract available. PMID 5818682
- [Background] Salmon SE, Haut A, Bonnet JD, Amare M, Weick JK, Durie BG, Dixon DO. Alternating combination chemotherapy and levamisole improves survival in multiple myeloma: a Southwest Oncology Group Study. J Clin Oncol. 1983 Aug;1(8):453-61. doi: 10.1200/JCO.1983.1.8.453. PMID 6366141
- [Background] Boccadoro M, Marmont F, Tribalto M, Avvisati G, Andriani A, Barbui T, Cantonetti M, Carotenuto M, Comotti B, Dammacco F, et al. Multiple myeloma: VMCP/VBAP alternating combination chemotherapy is not superior to melphalan and prednisone even in high-risk patients. J Clin Oncol. 1991 Mar;9(3):444-8. doi: 10.1200/JCO.1991.9.3.444. PMID 1999714
- [Background] MacLennan IC, Chapman C, Dunn J, Kelly K. Combined chemotherapy with ABCM versus melphalan for treatment of myelomatosis. The Medical Research Council Working Party for Leukaemia in Adults. Lancet. 1992 Jan 25;339(8787):200-5. doi: 10.1016/0140-6736(92)90004-m. PMID 1346171
- [Background] Blade J, San Miguel JF, Alcala A, Maldonado J, Sanz MA, Garcia-Conde J, Moro MJ, Alonso C, Besalduch J, Zubizarreta A, et al. Alternating combination VCMP/VBAP chemotherapy versus melphalan/prednisone in the treatment of multiple myeloma: a randomized multicentric study of 487 patients. J Clin Oncol. 1993 Jun;11(6):1165-71. doi: 10.1200/JCO.1993.11.6.1165. PMID 8501503
- [Background] Oken MM, Harrington DP, Abramson N, Kyle RA, Knospe W, Glick JH. Comparison of melphalan and prednisone with vincristine, carmustine, melphalan, cyclophosphamide, and prednisone in the treatment of multiple myeloma: results of Eastern Cooperative Oncology Group Study E2479. Cancer. 1997 Apr 15;79(8):1561-7. PMID 9118039
- [Background] Combination chemotherapy versus melphalan plus prednisone as treatment for multiple myeloma: an overview of 6,633 patients from 27 randomized trials. Myeloma Trialists' Collaborative Group. J Clin Oncol. 1998 Dec;16(12):3832-42. doi: 10.1200/JCO.1998.16.12.3832. PMID 9850028
- [Background] Gore ME, Selby PJ, Viner C, Clark PI, Meldrum M, Millar B, Bell J, Maitland JA, Milan S, Judson IR, et al. Intensive treatment of multiple myeloma and criteria for complete remission. Lancet. 1989 Oct 14;2(8668):879-82. doi: 10.1016/s0140-6736(89)91548-1. PMID 2571812
- [Background] Samson D, Gaminara E, Newland A, Van de Pette J, Kearney J, McCarthy D, Joyner M, Aston L, Mitchell T, Hamon M, et al. Infusion of vincristine and doxorubicin with oral dexamethasone as first-line therapy for multiple myeloma. Lancet. 1989 Oct 14;2(8668):882-5. doi: 10.1016/s0140-6736(89)91549-3. PMID 2571813
- [Background] Hjorth M, Holmberg E, Rodjer S, Turesson I, Westin J, Wisloff F. Survival in conventionally treated younger (<60 years) multiple myeloma patients: no improvement during two decades. Nordic Myeloma Study Group (NMSG). Eur J Haematol. 1999 Apr;62(4):271-7. doi: 10.1111/j.1600-0609.1999.tb01757.x. PMID 10227461
- [Background] Lokhorst HM, Schattenberg A, Cornelissen JJ, Thomas LL, Verdonck LF. Donor leukocyte infusions are effective in relapsed multiple myeloma after allogeneic bone marrow transplantation. Blood. 1997 Nov 15;90(10):4206-11. PMID 9354693
- [Background] Gahrton G, Tura S, Ljungman P, Blade J, Brandt L, Cavo M, Facon T, Gratwohl A, Hagenbeek A, Jacobs P, et al. Prognostic factors in allogeneic bone marrow transplantation for multiple myeloma. J Clin Oncol. 1995 Jun;13(6):1312-22. doi: 10.1200/JCO.1995.13.6.1312. PMID 7751876
- [Background] Bensinger WI, Buckner CD, Anasetti C, Clift R, Storb R, Barnett T, Chauncey T, Shulman H, Appelbaum FR. Allogeneic marrow transplantation for multiple myeloma: an analysis of risk factors on outcome. Blood. 1996 Oct 1;88(7):2787-93. PMID 8839877
- [Background] Powles R, Raje N, Milan S, Millar B, Shepherd V, Mehta J, Singhal S, Kulkarni S, Viner C, Gore M, Cunningham D, Treleaven J. Outcome assessment of a population-based group of 195 unselected myeloma patients under 70 years of age offered intensive treatment. Bone Marrow Transplant. 1997 Sep;20(6):435-43. doi: 10.1038/sj.bmt.1700917. PMID 9313875
- [Background] Vesole DH, Tricot G, Jagannath S, Desikan KR, Siegel D, Bracy D, Miller L, Cheson B, Crowley J, Barlogie B. Autotransplants in multiple myeloma: what have we learned? Blood. 1996 Aug 1;88(3):838-47. PMID 8704239
- [Background] Barlogie B, Jagannath S, Naucke S, Mattox S, Bracy D, Crowley J, Tricot G, Alexanian R. Long-term follow-up after high-dose therapy for high-risk multiple myeloma. Bone Marrow Transplant. 1998 Jun;21(11):1101-7. doi: 10.1038/sj.bmt.1701182. PMID 9645572
- [Background] 23. Barlogie B, Ayers D, Spoon D, et al. Towards curing myeloma. durable CR in the absence of chromosome 13 deletion and with timely application of two cycles of melphalan-based high dose therapy. Proceedings of the VII International Multiple Myeloma Workshop, Stockholm, September 1999, pp: 49.
- [Background] Alexanian R, Weber D, Delasalle K, Dimopoulos M, Giralt S, Champlin R. Early myeloablative therapy with autologous stem cells for multiple myeloma in remission with primary therapy. Proceedings of the VII International Multiple Myeloma Workshop, Stockholm, September 1999, pp: 61.
- [Background] 25. Bladé J, Esteve J, Rives S, et al. Early autologous stem cell transplantation versus standard chemotherapy after first response in multipple myeloma: a report of a non-randomized study from a single institution. Proceedings of the VII International Multiple Myeloma Workshop, Stockholm, September 1999, pp: 148.
- [Background] Lahuerta JJ, Martinez-Lopez J, Serna JD, Blade J, Grande C, Alegre A, Vazquez L, Garcia-Larana J, Sureda A, Rubia JD, Conde E, Martinez R, Perez-Equiza K, Moraleda JM, Leon A, Besalduch J, Cabrera R, Miguel JD, Morales A, Garcia-Ruiz JC, Diaz-Mediavilla J, San-Miguel J. Remission status defined by immunofixation vs. electrophoresis after autologous transplantation has a major impact on the outcome of multiple myeloma patients. Br J Haematol. 2000 May;109(2):438-46. doi: 10.1046/j.1365-2141.2000.02012.x. PMID 10848839
- [Background] Attal M, Harousseau JL, Stoppa AM, Sotto JJ, Fuzibet JG, Rossi JF, Casassus P, Maisonneuve H, Facon T, Ifrah N, Payen C, Bataille R. A prospective, randomized trial of autologous bone marrow transplantation and chemotherapy in multiple myeloma. Intergroupe Francais du Myelome. N Engl J Med. 1996 Jul 11;335(2):91-7. doi: 10.1056/NEJM199607113350204. PMID 8649495
- [Background] Palumbo A, Triolo S, Argentino C, Bringhen S, Dominietto A, Rus C, Omede P, Tarella C, Pileri A, Boccadoro M. Dose-intensive melphalan with stem cell support (MEL100) is superior to standard treatment in elderly myeloma patients. Blood. 1999 Aug 15;94(4):1248-53. PMID 10438712
- [Background] Barlogie B, Jagannath S, Vesole DH, Naucke S, Cheson B, Mattox S, Bracy D, Salmon S, Jacobson J, Crowley J, Tricot G. Superiority of tandem autologous transplantation over standard therapy for previously untreated multiple myeloma. Blood. 1997 Feb 1;89(3):789-93. PMID 9028309
- [Background] Lenhoff S, Hjorth M, Holmberg E, Turesson I, Westin J, Nielsen JL, Wisloff F, Brinch L, Carlson K, Carlsson M, Dahl IM, Gimsing P, Hippe E, Johnsen HE, Lamvik J, Lofvenberg E, Nesthus I, Rodjer S. Impact on survival of high-dose therapy with autologous stem cell support in patients younger than 60 years with newly diagnosed multiple myeloma: a population-based study. Nordic Myeloma Study Group. Blood. 2000 Jan 1;95(1):7-11. PMID 10607678
- [Background] Blade J, San Miguel JF, Fontanillas M, Alcala A, Maldonado J, Garcia-Conde J, Conde E, Conzalez-Brito G, Moro MJ, Escudero ML, Trujillo J, Pascual A, Rozman C, Estape J, Montserrat E. Survival of multiple myeloma patients who are potential candidates for early high-dose therapy intensification/ autotransplantation and who were conventionally treated. J Clin Oncol. 1996 Jul;14(7):2167-73. doi: 10.1200/JCO.1996.14.7.2167. PMID 8683251
- [Background] Alexanian R, Dimopoulos MA, Hester J, Delasalle K, Champlin R. Early myeloablative therapy for multiple myeloma. Blood. 1994 Dec 15;84(12):4278-82. PMID 7994043
- [Background] Vesole DH, Barlogie B, Jagannath S, Cheson B, Tricot G, Alexanian R, Crowley J. High-dose therapy for refractory multiple myeloma: improved prognosis with better supportive care and double transplants. Blood. 1994 Aug 1;84(3):950-6. PMID 7913845
- [Background] Singhal S, Mehta J, Desikan R, Ayers D, Roberson P, Eddlemon P, Munshi N, Anaissie E, Wilson C, Dhodapkar M, Zeddis J, Barlogie B. Antitumor activity of thalidomide in refractory multiple myeloma. N Engl J Med. 1999 Nov 18;341(21):1565-71. doi: 10.1056/NEJM199911183412102. PMID 10564685
- [Background] 35. Singhal S, Mehta J., Eddlemon P., Gray P., Cromer J., Desikan R., Ayers D., Siegel D., Munshi N., Anaissie E., Kantarjian H., Zeldis J., Barlogie B. Marked anti-tumor effect from anti-angiogenesis therapy with thalidomide in high risk refractory multiple myeloma. Blood, 1998; 92(suppl 1):318a (abstract).
- [Background] Rajkumar SV, Hayman S, Gertz MA, Dispenzieri A, Lacy MQ, Greipp PR, Geyer S, Iturria N, Fonseca R, Lust JA, Kyle RA, Witzig TE. Combination therapy with thalidomide plus dexamethasone for newly diagnosed myeloma. J Clin Oncol. 2002 Nov 1;20(21):4319-23. doi: 10.1200/JCO.2002.02.116. PMID 12409330
- [Background] Weber D, Rankin K, Gavino M, Delasalle K, Alexanian R. Thalidomide alone or with dexamethasone for previously untreated multiple myeloma. J Clin Oncol. 2003 Jan 1;21(1):16-9. doi: 10.1200/JCO.2003.03.139. PMID 12506164
- [Background] 38. Rajkumar S, Blood E, Vesole D, Shepard R, Greipp P. Thalidomide plus dexamethasone versus dexamethasone alone in newly diagnosed multiple myeloma. Blood 2004. Volume 104, issue 11. Abstract 205
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] Jagannath S, Barlogie B, Berenson J, Siegel D, Irwin D, Richardson PG, Niesvizky R, Alexanian R, Limentani SA, Alsina M, Adams J, Kauffman M, Esseltine DL, Schenkein DP, Anderson KC. A phase 2 study of two doses of bortezomib in relapsed or refractory myeloma. Br J Haematol. 2004 Oct;127(2):165-72. doi: 10.1111/j.1365-2141.2004.05188.x. PMID 15461622
- [Background] 41. Paul Richardson et al. Bortezomib Demonstrates Superior Efficacy to High-Dose Dexamethasone in Relapsed Multiple Myeloma: Final Report of the APEX Study. Blood 2004; 104(11):Abstract number 336.5
- [Background] 42. Maurizio Zangari, Bart Barlogie, Joth Jacobson, Erik Rasmussen, Michael Burns, Bob Kordsmeier, John D. Shaughnessy, Elias J. Anaissie, Raymond Thertulien, Athanasios Fassas, Choon-Kee Lee, David Schenkein, Jerome B. Zeldis, Guido Tricot. VTD Regimen Comprising Velcade (V) + Thalidomide (T) and Added DEX (D) for Non-Responders to V + T Effects a 57% PR Rate among 56 Patients with Myeloma (M) Relapsing after Autologous Transplant. Blood 2003, Volume 102, issue 11. Abstract number 830
- [Background] 43. Jagannath S, Brian D, Wolf j, Camacho E, Irwin D, Lutzky J, Mckinley M, Gabayan E, Mazumder A, Crowley K, Sckenkein D. A phase 2 study of Bortezomib as first-line therapy in patients with multiple myeloma. Blood 2004; 104(11). Abstract number 333
- [Background] 44. Alexanian R, Wang L, Weber D, Delasalle K. VTD (Velcade, Thalidomide, Dexamethasone) as primary therapy for newly-diagnosed multiple myeloma. Blood 2004; 104(11). Abstract number 210
- [Background] Desikan KR, Barlogie B, Jagannath S, Vesole DH, Siegel D, Fassas A, Munshi N, Singhal S, Mehta J, Tindle S, Nelson J, Bracy D, Mattox S, Tricot G. Comparable engraftment kinetics following peripheral-blood stem-cell infusion mobilized with granulocyte colony-stimulating factor with or without cyclophosphamide in multiple myeloma. J Clin Oncol. 1998 Apr;16(4):1547-53. doi: 10.1200/JCO.1998.16.4.1547. PMID 9552064
- [Background] 46. Whealthy K (On behalf of the Myeloma Trialists'Collaborative Group). Which myeloma patients benefit from interferon therapy? An overview of 24 randomised trials with 4,000 patients, Br J Haematol 1998; 102: 140.
- [Background] Blade J, Esteve J. Viewpoint on the impact of interferon in the treatment of multiple myeloma: benefit for a small proportion of patients? Med Oncol. 2000 May;17(2):77-84. doi: 10.1007/BF02796202. PMID 10871813
- [Background] Palumbo A, Boccadoro M, Garino LA, Gallone G, Frieri R, Pileri A. Multiple myeloma: intensified maintenance therapy with recombinant interferon-alpha-2b plus glucocorticoids. Eur J Haematol. 1992 Aug;49(2):93-7. doi: 10.1111/j.1600-0609.1992.tb00037.x. PMID 1397246
- [Background] Salmon SE, Crowley JJ, Balcerzak SP, Roach RW, Taylor SA, Rivkin SE, Samlowski W. Interferon versus interferon plus prednisone remission maintenance therapy for multiple myeloma: a Southwest Oncology Group Study. J Clin Oncol. 1998 Mar;16(3):890-6. doi: 10.1200/JCO.1998.16.3.890. PMID 9508170
- [Background] Berenson JR, Crowley JJ, Grogan TM, Zangmeister J, Briggs AD, Mills GM, Barlogie B, Salmon SE. Maintenance therapy with alternate-day prednisone improves survival in multiple myeloma patients. Blood. 2002 May 1;99(9):3163-8. doi: 10.1182/blood.v99.9.3163. PMID 11964279
- [Background] International Myeloma Working Group. Criteria for the classification of monoclonal gammopathies, multiple myeloma and related disorders: a report of the International Myeloma Working Group. Br J Haematol. 2003 Jun;121(5):749-57. PMID 12780789
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- [Background] Rizzo JD, Lichtin AE, Woolf SH, Seidenfeld J, Bennett CL, Cella D, Djulbegovic B, Goode MJ, Jakubowski AA, Lee SJ, Miller CB, Rarick MU, Regan DH, Browman GP, Gordon MS; American Society of Clinical Oncology; Americcan Society of Hematology. Use of epoetin in patients with cancer: evidence-based clinical practice guidelines of the American Society of Clinical Oncology and the American Society of Hematology. Blood. 2002 Oct 1;100(7):2303-20. doi: 10.1182/blood-2002-06-1767. PMID 12239138
- [Background] Rizzo JD, Lichtin AE, Woolf SH, Seidenfeld J, Bennett CL, Cella D, Djulbegovic B, Goode MJ, Jakubowski AA, Lee SJ, Miller CB, Rarick MU, Regan DH, Browman GP, Gordon MS; American Society of Clinical Oncology. American Society of Hematology. Use of epoetin in patients with cancer: evidence-based clinical practice guidelines of the American Society of Clinical Oncology and the American Society of Hematology. J Clin Oncol. 2002 Oct 1;20(19):4083-107. doi: 10.1200/JCO.2002.07.177. PMID 12351606
- [Derived] Rosinol L, Hebraud B, Oriol A, Colin AL, Rios Tamayo R, Hulin C, Blanchard MJ, Caillot D, Sureda A, Hernandez MT, Arnulf B, Mateos MV, Macro M, San-Miguel J, Belhadj K, Lahuerta JJ, Garelik MB, Blade J, Moreau P. Integrated analysis of randomized controlled trials evaluating bortezomib + lenalidomide + dexamethasone or bortezomib + thalidomide + dexamethasone induction in transplant-eligible newly diagnosed multiple myeloma. Front Oncol. 2023 Nov 2;13:1197340. doi: 10.3389/fonc.2023.1197340. eCollection 2023. PMID 38023148
- [Derived] Sonneveld P, Goldschmidt H, Rosinol L, Blade J, Lahuerta JJ, Cavo M, Tacchetti P, Zamagni E, Attal M, Lokhorst HM, Desai A, Cakana A, Liu K, van de Velde H, Esseltine DL, Moreau P. Bortezomib-based versus nonbortezomib-based induction treatment before autologous stem-cell transplantation in patients with previously untreated multiple myeloma: a meta-analysis of phase III randomized, controlled trials. J Clin Oncol. 2013 Sep 10;31(26):3279-87. doi: 10.1200/JCO.2012.48.4626. Epub 2013 Jul 29. PMID 23897961
- [Derived] Rosinol L, Oriol A, Teruel AI, Hernandez D, Lopez-Jimenez J, de la Rubia J, Granell M, Besalduch J, Palomera L, Gonzalez Y, Etxebeste MA, Diaz-Mediavilla J, Hernandez MT, de Arriba F, Gutierrez NC, Martin-Ramos ML, Cibeira MT, Mateos MV, Martinez J, Alegre A, Lahuerta JJ, San Miguel J, Blade J; Programa para el Estudio y la Terapeutica de las Hemopatias Malignas/Grupo Espanol de Mieloma (PETHEMA/GEM) group. Superiority of bortezomib, thalidomide, and dexamethasone (VTD) as induction pretransplantation therapy in multiple myeloma: a randomized phase 3 PETHEMA/GEM study. Blood. 2012 Aug 23;120(8):1589-96. doi: 10.1182/blood-2012-02-408922. Epub 2012 Jul 12. PMID 22791289
- [Derived] Sarasquete ME, Gutierrez NC, Misiewicz-Krzeminska I, Paiva B, Chillon MC, Alcoceba M, Garcia-Sanz R, Hernandez JM, Gonzalez M, San-Miguel JF. Upregulation of Dicer is more frequent in monoclonal gammopathies of undetermined significance than in multiple myeloma patients and is associated with longer survival in symptomatic myeloma patients. Haematologica. 2011 Mar;96(3):468-71. doi: 10.3324/haematol.2010.033845. Epub 2010 Dec 15. PMID 21160068
- See also: Spanish association of Haematology — http://www.aehh.org